CLINICAL TRIAL: NCT05977361
Title: Intrathecal Catheter Placement Versus Resiting Epidural Catheter After Dural Puncture in Obstetric Patients: a Multicenter Randomized Controlled Trial
Brief Title: Intrathecal Catheter Placement Versus Resiting Epidural Catheter After Dural Puncture in Obstetric Patients
Acronym: ItaREVI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ItaREVI
Record Dates: First submitted 2023-07-20; First posted 2023-08-04 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2023-07

CONDITIONS: Analgesia, Obstetrical; Post-Dural Puncture Headache
Keywords: Labor Pain; Obstetric Labor Complications; Analgesia, Epidural
MeSH Terms: conditions — Agnosia; Post-Dural Puncture Headache; Labor Pain; Obstetric Labor Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resiting Epidural Catheter (Active Comparator)
  Interventions: Procedure: Resiting Epidural Catheter
- Intrathecal catheter placement (Active Comparator)
  Interventions: Procedure: Intrathecal Catheter Placement

INTERVENTIONS:
Procedure: Resiting Epidural Catheter — After a UDP has occurred, epidural catheter will be re-sited in a different intervertebral space. Analgesia will be then maintained according to internal protocol, using PIEB (Programmed Intermittent Epidural Bolus) system. Catheter will be left in place for the first 24-36 hours.
  Arms: Resiting Epidural Catheter
Procedure: Intrathecal Catheter Placement — After a UDP has occurred, an intrathecal catheter will be placed through the dural tap. Analgesia will be then maintained according to internal protocol, using PISB (Programmed Intermittent Subarachnoid Bolus) system. Catheter will be left in place for the first 24-36 hours. During this time, a continuous infusion of sterile saline at a rate of 2 mL/h will be maintained. Before removal, an additional bolus of 10 mL of sterile saline will be administered in the intrathecal catheter.
  Arms: Intrathecal catheter placement

SUMMARY:
Epidural anesthesia represents the most popular method for pain relief during labour. Unintentional dural puncture (UDP) occurs in 0.4-1.5% of labour epidural analgesia, representing therefore the most common complication. Up to 80% of patients with a UDP may develop a post-dural puncture headache (PDPH).

When a UDP occurs, two possible strategies have been proposed in order to ensure analgesia during labour: either resiting the epidural catheter in a different intervertebral space, or inserting an intrathecal catheter. Both strategies proved to equally provide analgesia during labour, but their relative contribution in preventing PDPH is still not known.

The primary aim of this multicenter randomized controlled trial is therefore to compare these two strategies in the occurrence of PDPH at 24 hours from the UDP.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of UDP during labour
* Written informed consent

Exclusion Criteria:

* Refusal to participate in the study
* History of PDPH

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Estimated)
Dates: Start 2024-04-26 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
PDPH incidence | At 24 hours from UDP
  Incidence of post-dural puncture headache (PDPH) at 24 hours from UDP occurrence

SECONDARY OUTCOMES:
PDPH intensity at 24 hours | At 24 hours from UDP
  PDPH intensity, rated using a 10-point scale, ranging from 0 ("no pain") to 10 ("worst pain imaginable")
PDPH intensity at 48 hours | At 48 hours from UDP
  PDPH intensity, rated using a 10-point scale, ranging from 0 ("no pain") to 10 ("worst pain imaginable")
Quality of analgesia | During the entire course of labour, an average of 12 hours
  Quality of analgesia during labour will be evaluated, based on the number of additional boluses of local anesthetic administered during labour to treat breakthrough pain.
Adverse events | During the entire follow-up period, up to 3 months from UDP
  All reported adverse events, including number of unsuccessful attempts at placing the epidural or subarachnoid catheter, motor block, poor analgesia, caesarean section rate.
Chronic pain at 1 month | At 1 month from UDP
  Incidence of chronic headache and chronic low back pain
Chronic pain at 3 months | At 3 months from UDP
  Incidence of chronic headache and chronic low back pain
Readmission to hospital | Up to 3 months from UDP
  ER visits or hospital readmissions due to neurological symptoms related or possibly related to PDPH (severe headache, severe back pain, fever, leg weakness, incontinence of urine or stool)
Patient's satisfaction | Before discharge, an average of 1 week
  Patient's satisfaction, evaluated through the Italian version of the Birth Satisfaction Scale-Revised (BSS-R)

IPD SHARING:
Plan to Share IPD: No